CLINICAL TRIAL: NCT04876326
Title: Potential Use of Autologous and Allogeneic Mesenchymal Stem Cells in Patients With Multiple System Atrophy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Ismail Hadisoebroto Dilogo, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TGHISMMSCMSA
Record Dates: First submitted 2021-04-25; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Multiple System Atrophy; Parkinsonism; Multiple System Atrophy, Parkinson Variant
Keywords: Multiple System Atrophy, Parkinson Variant; Mesenchymal Stem Cell; Parkinsonism; UMSARS; MRI; FGD-PET SCAN; DaTScan; SSR, RR-Interval; Composite Autonomic Severity Score; ILG-1, BDNF; ERG (Electroretinogram); VEP (Visual Evoked Potential); HD-OCT (High Definition-optical coherence tomography)
MeSH Terms: conditions — Multiple System Atrophy; Parkinsonian Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Autologous Adipose MSC Group (Active Comparator): This group will receive the implantation of autologous mesenchymal stem cell origin of adipose tissue with a dose of 2 x 50 million cells given with a distance of 1 month
  Interventions: Biological: Autologous Adipose Mesenchymal Stem Cell Implantation
- Allogeneic Umbilical Cord MSC Group (Active Comparator): This group will receive intrathecal implantation of allogeneic mesenchymal stem cells from the umbilical cord with a dose of 2 x 50 million cells given a distance of 1 month.
  Interventions: Biological: Allogeneic Umbilical Cord Mesenchymal Stem Cell Implantation
- Allogeneic Umbilical Cord MSC and Adipose Secretome Group (Active Comparator): This group will receive intrathecal implantation of allogeneic mesenchymal stem cells from the umbilical cord as much as 2 x 50 million followed by 2 x 10cc mesenchymal stem cell secretions from adipose tissue intravenously given at a distance of 1 month.
  Interventions: Biological: Allogeneic Umbilical Cord Mesenchymal Stem Cell and Adipose Secretome Implantation

INTERVENTIONS:
Biological: Autologous Adipose Mesenchymal Stem Cell Implantation — Before taking adipose tissue, each subject was screened including HbSAg, Anti HbS, Anti HCV, HIC, MCV and syphilis tests.
  Adipose tissue was taken through 5 grams of subcutaneous fat biopsy from the abdomen of each subject and put into a transport medium and then sent to the RSCM-FKUI cGMP IPT Stem Cells Laboratory for immediate isolation of mesenchymal stem cells.
  MSC that has been isolated will be cultured using the appropriate medium until it reaches the desired passage and the number of cells.
  The viability and proliferation ability of cultured cells were evaluated, then characterization of cell antigen expression was carried out using flow cytometry to confirm the success of MSC culture.
  The MSC to be injected into the subject will be prepared in 2cc physiological NaCl transport medium just before implantation.
  The adipose secretion used is prepared in whole form as much as 10cc in a 10cc syringe.
  Arms: Autologous Adipose MSC Group
Biological: Allogeneic Umbilical Cord Mesenchymal Stem Cell Implantation — Before taking the umbilical cord tissue, a pregnant woman's donor was screened including HbSAg, Anti HbS, Anti HCV, HIC, MCV and syphilis tests.
  Immediately after delivery, the umbilical cord was collected and stored in a sterile specimen plate containing 0.9% NaCl at 4⁰C.
  The umbilical cord is transported to the GMP standard culture laboratory at the UPT TK Stem Cells RSCM-FKUI for isolation process of mesenchymal stem cells. Sample processing was carried out within 8 hours of delivery to maintain cell viability.
  MSC that has been isolated will be cultured using the appropriate medium until it reaches the desired passage and the number of cells.
  The viability and proliferation ability of cultured cells were evaluated, then characterization of cell antigen expression was carried out using flow cytometry to confirm the success of MSC culture.
  The MSC to be injected into the subject will be prepared in a suitable transport medium just prior to implantation.
  Arms: Allogeneic Umbilical Cord MSC Group
Biological: Allogeneic Umbilical Cord Mesenchymal Stem Cell and Adipose Secretome Implantation — Before taking adipose and umbilical cord tissue, each subject was screened. -For Adipose tissue : The adipose secretion used is prepared in whole form as much as 10cc in a 10cc syringe.
  -Uc-MSC : Immediately after delivery, the umbilical cord was collected and stored in a sterile specimen plate containing 0.9% NaCl at 4⁰C.
  The umbilical cord is transported to the GMP standard culture laboratory to have isolation process of mesenchymal stem cells. Sample processing was carried out within 8 hours of delivery to maintain cell viability.
  Later it will be cultured using the appropriate medium until it reaches the desired passage and the number of cells.The viability and proliferation ability of cultured cells were evaluated, then characterization of cell antigen expression was carried out using flow cytometry to confirm the success of MSC culture.
  Arms: Allogeneic Umbilical Cord MSC and Adipose Secretome Group

SUMMARY:
The prevalence of Multiple System Atrophy (MSA) is reported to be between 3.4 - 4.9 cases per 100,000 population. The estimated average incidence is 0.6 - 0.7 cases per 100,000 people per year. Many patients are not diagnosed properly during their lifetime because of the difficulty in differentiating MSA from other disorders. Approximately 29 - 33% of patients with isolated late onset cerebellar ataxia and 8 - 10% of patients with parkinsonism will develop MSA.

There are currently no therapies that can cure or stop the progression of the disease. The current pharmacological therapy is only to relieve symptoms. Mesenchymal stem cells (MSC) are considered an efficient source of cells for therapy, because they can be safely harvested and transplanted to donors or patients, have low immunogenicity, and have broad therapeutic potential. Results from preliminary preclinical and clinical trials indicate the potential of MSC-based treatment in meeting several key aspects of neurodegeneration. Stem cell-based therapy for neurodegenerative diseases aims to stop clinical damage by regenerating and by providing local support for damaged tissue, in addition after transplantation, MSCs have been shown to be capable of penetrating the lesion area and thus have great potential use as a means of administering therapeutic agents.

The subjects of this study were patients who experienced possible MSA based on the consensus clinical criteria for MSA. There will be three treatment groups with a total sample of 5 subjects each.

Group 1 will receives MSC-Adipose Autologous with doses 2x50 million cells intratechally.

Group 2 will receives MSC-Umbilical Cord Allogeneic with doses 2x 50 million cells intratechally.

Group 3 will receives MSC-Umbilical Cord Allogeneic with doses 2x50 million cells intratechally and 2x10cc secretome MSC from Adipose Intravenously.

Clinical improvement will be evaluated using the UMSARS scale, PET-Scans, MRI, DaTScan, IGF-1, BDNF, Sympathetic skin respons (SSR), EMG, Composite Autonomic Severity Score (CASS), High definition-Optical coherence tomography (HD-OCT), ERG, VEP, Log MAR chart, Ishihara test and side adverse effect on MSC.

This study is divided into six timeframes : Before an implantation, First Month after second implantation, Third month after secondary implantation, Sixth month after second implantation, Ninth month after second implantation and Twelve month after second implantation. The differences between the test variables are then used as an indicator to assess clinical improvement within the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients developed MSA based on clinical examination and consensus MSA criteria.
* Patients diagnosed with MSA for less than 4 years.
* Patients with an anticipated survival of at least 3 years in the opinion of the examiner.
* Patients with MOCa and Mini Mental State Examination (MMSE) values of more than 24.
* For Adipose Autologous-MSC group subjects were not experiencing active infection, which was confirmed by screening for HbSAg, Anti HCV, Syphilis, HIV, CMV, Rubella, and Toxoplasma.
* Subjects are willing to participate in research and fill out an informed consent form.
* Do not have autoimmune disorder, or undergoes management disorders and / or other diseases related to MSA
* Subjects are willing to participate in research and fill out an informed consent form.

Exclusion Criteria:

* Suffer from systemic autoimmune diseases (systemetic lupus erythomatosus, Addison's disease, Crohn's disease, arthritis management), immunodeficiency (SIDA), or blood clotting disorders or management of malignant diseases (diseases associated with MSA)
* Undergo immunosuppressive therapy, anticoagulants or corticosteroids.
* Patients with malignant neoplasms and close family history of neoplasms.
* already had history of spinal surgery, have paralysis or have spinal diseases.
* Patients with a history of electroconvulsive therapy.
* Patients with a history of brain surgery for Parkinson's disease.
* Patients with systemic or local infections located close to the injection site.
* Undergo immunosuppressive therapy, anticoagulants or corticosteroids.
* The patient was not willing to take part in the study and did not fill out informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-10-05 (Estimated); Study Completion 2021-10-05 (Estimated)

PRIMARY OUTCOMES:
Changes of Clinical Evaluation from Baseline to 1,3,6,9 and 12 months after second implantation | Pre-implantation, 1st Month, 3rd Months, 6th Months , 9th, 12th Months After Second Implantation
  Subjects will be evaluated by Neurological test
Changes of Clinical Evaluation from Baseline to 1,3,6,9 and 12 months after second implantation | Pre-implantation, 1st Month, 3rd Months, 6th Months , 9th, 12th Months After Second Implantation
  Subjects will be evaluated by UMSARS(Unified Multiple System Atrophy Rating Scale)
Changes of structures improvement of the eyes from Baseline to 1,3,6,9 and 12 months after second implantation | Pre-implantation, 1st Month, 3rd Months, 6th Months , 9th, 12th Months After Second Implantation
  an increase in the thickness of the Retinal Nerve Fiber Layer(RNFL) checked from the High Definition-Optical Coherence Tomography examination(HD-OCT)
Changes of structures improvement of the eyes from Baseline to 1,3,6,9 and 12 months after second implantation | Pre-implantation, 1st Month, 3rd Months, 6th Months , 9th, 12th Months After Second Implantation
  an increase in the Ganglion Cell Complex (GCC) checked from the High Definition-Optical Coherence Tomography examination(HD-OCT)
Changes of the eyesight from Baseline to 1,3,6,9 and 12 months after second implantation | Pre-implantation, 1st Month, 3rd Months, 6th Months , 9th, 12th Months After Second Implantation
  improvement of eyesight will be checked using LogMar Test
Changes of the eyesight from Baseline to 1,3,6,9 and 12 months after second implantation | Pre-implantation, 1st Month, 3rd Months, 6th Months , 9th, 12th Months After Second Implantation
  improvement of eyesight will be checked using Ishihara test
Changes of the eyesight from Baseline to 1,3,6,9 and 12 months after second implantation | Pre-implantation, 1st Month, 3rd Months, 6th Months , 9th, 12th Months After Second Implantation
  improvement of eyesight will be checked using VEP (Visual Evoked Potential)
Changes of the eyesight from Baseline to 1,3,6,9 and 12 months after second implantation | Pre-implantation, 1st Month, 3rd Months, 6th Months , 9th, 12th Months After Second Implantation
  improvement of eyesight will be checked using ERG (Electroretinogram)
Imaging Evaluation from Baseline to 1,3,6,9 and 12 months after second implantation | Pre-implantation, 1st Month, 3rd Months, 6th Months , 9th, 12th Months After Second Implantation
  The Brain will be checked to see Changes of MRI to see increased FDG Uptake
Imaging Evaluation from Baseline to 1,3,6,9 and 12 months after second implantation | Pre-implantation, 1st Month, 3rd Months, 6th Months , 9th, 12th Months After Second Implantation
  The Brain will be checked to see Changes of FGD-PET SCAN to see increased FDG Uptake
Imaging Evaluation from Baseline to 1,3,6,9 and 12 months after second implantation | Pre-implantation, 1st Month, 3rd Months, 6th Months , 9th, 12th Months After Second Implantation
  The Brain will be checked to see Changes of DaTScan to see increased FDG Uptake

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo General Hospital, Jakarta Pusat, DKI Jakarta, Indonesia